CLINICAL TRIAL: NCT02935179
Title: Office of Human Research, Taipei Medical University
Brief Title: The Effect of White Sweet Potato Meal Replacement on Weight Control of the Obesity
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Taipei Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: N201604045
Record Dates: First submitted 2016-10-14; First posted 2016-10-17 (Estimated); Results first posted 2019-04-17 (Actual); Last update posted 2019-04-30 (Actual); Status verified 2016-06

CONDITIONS: Overweight
MeSH Terms: conditions — Overweight

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Control Group (Placebo Comparator): Normal diet with 1500~2000 kcal
  Interventions: Dietary Supplement: White sweet potato diet
- Treatment Group (Experimental): White sweet potato diet with 1500~2000 kcal
  Interventions: Dietary Supplement: White sweet potato diet

INTERVENTIONS:
Dietary Supplement: White sweet potato diet — The diet were supplied 516 kcal daily

SUMMARY:
The purpose of this project is to use white-skinned sweet potato as the main material for weight control for overweight and obesity, the non-communicable diseases (cardiovascular diseases, cancers, chronic respiratory diseases and diabetes) are also included. All high quality sweet potato are provided by CAES in Taiwan to produce special nutrient food and health food that to do functional study in Shih Chien University and Taipei Medical University. In this study, the investigators will recruit overweight and obesity subjects that divide into white sweet potato group (experimental group) and no intervention group (control group) by using randomized, parallel and open clinical study in sixty days.

DETAILED DESCRIPTION:
All subjects will be evaluated the body weight and clinical nutrition assessment such as postural measurement, urine test and blood biomarker examination.

ELIGIBILITY:
Inclusion Criteria:

* 24≦ BMI≦30

Exclusion Criteria:

* Pregnant and lactating women
* Patients within six months after surgery
* Mental illness or depression
* Suffering from cancer, ulcers, acute respiratory infections, dialysis, acute hepatitis and other diseases
* Those who have taken "additional nutritional supplements" habit

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2016-07; Primary Completion 2016-12 (Actual); Study Completion 2017-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Chih-Han Lin, MS, Principal Investigator — Office of Human Research, Taipei Medical University

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Control Group: Normal diet
  White sweet potato meal replacement: The formula were supplied 516 kcal daily
- Treatment Group: Normal diet plus white sweet potato formula
  White sweet potato meal replacement: The formula were supplied 516 kcal daily
Period: Overall Study
Arm/Group | Control Group | Treatment Group
Started | 30 | 30
Completed | 29 | 29
Not Completed | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Control Group | Treatment Group | Total
Number analyzed (Participants) | 29 | 29 | 58
Age, Continuous [Mean (Standard Deviation); unit: years] | 37.33 (5.51) | 38.76 (6.24) | 38.07 (5.89)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14 | 14 | 28
  Male | 15 | 15 | 30

OUTCOME MEASURES:

1. Primary Outcome: Body Weight After Intervention
Description: Body weight change after 60 days intervention
Time Frame: 60 days
Measure: Mean (Standard Deviation); unit: Kg
Arm/Group | Control Group | Treatment Group
Number analyzed (Participants) | 29 | 29
Kg | -2.11 (1.7) | -3.7 (2.24)

2. Secondary Outcome: Body Fat After Intervention
Description: Body fat change after 60 days intervention
Time Frame: 60 days
Measure: Mean (Standard Deviation); unit: percentage of body fat
Arm/Group | Control Group | Treatment Group
Number analyzed (Participants) | 29 | 29
percentage of body fat | -0.95 (2.21) | -2.26 (2.09)

ADVERSE EVENTS:
Time Frame: The adverse event data were collected from the participants during intervention and assessed after 24 weeks.
Description: No adverse event.
Arm/Group | Control Group | Treatment Group
All-Cause Mortality (participants affected / at risk) | 0/29 | 0/29
Serious Adverse Events (participants affected / at risk) | 0/29 | 0/29
Other Adverse Events (participants affected / at risk) | 0/29 | 0/29

LIMITATIONS AND CAVEATS:
Small sample size and trial duration that may cause impose an obstacle in the detection of significant changes of the study measure.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No